CLINICAL TRIAL: NCT05613062
Title: A Randomized Placebo-Controlled Pilot Study of an Herbal Formula Modified Huang-Lian-Jie-Du Decoction (MHLJDD) for Atopic Dermatitis in Children
Brief Title: Modified Huang-Lian-Jie-Du Decoction (MHLJDD) for Atopic Dermatitis in Children
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD HLJDD study
Record Dates: First submitted 2022-09-29; First posted 2022-11-14 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Modified Huang-Lian-Jie-Du Decoction (MHLJDD)) (Experimental): Chinese medicine
  Interventions: Drug: Modified Huang-Lian-Jie-Du Decoction (MHLJDD)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modified Huang-Lian-Jie-Du Decoction (MHLJDD) — Chinese medicine granules for 12 weeks twice daily
  Other Names: Chinese medicine
  Arms: Active treatment (Modified Huang-Lian-Jie-Du Decoction (MHLJDD))
Drug: Placebo — Placebo granules for 12 weeks twice daily
  Arms: Placebo

SUMMARY:
The study aims to evaluate the clinical efficacy of Chinese medicine (CM) for the treatment of subacute and chronic Atopic Dermatitis (AD) patients when compared to the placebo control by examining the clinical symptoms.

DETAILED DESCRIPTION:
This is a parallel, randomized, placebo-controlled, double-blind pilot study. The subjects will come for a screening visit at week 0 (baseline), then at week 6±3 days, week 12±3 days and week 16±4 days for Chinese medicine practitioner (CMP) investigators' assessments (Fig 1). Eczema Area and Severity Index (EASI), Children's dermatology life quality index (CDLQI), and Patient-Oriented Eczema Measure (POEM) will be assessed and filled up at different time points. Eligible subjects will be randomly allocated to the treatment group receiving oral CM granules or the placebo control group receiving oral placebo granules for 12 weeks, and then be followed up 4 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age of 4 to 17 (Chinese only);
* With EASI ≥ 10;
* Subacute and chronic atopic dermatitis presenting with dry, scaly, erythematous papules and plaques; and
* Provide a written informed consent form (signed by one of their parents)

Exclusion Criteria:

* History of allergy to Chinese medicines;
* AD with Yang deficiency in syndrome differentiation, such as pale looking, always feeling cold, fatigue, chronic diarrhea with loose stool, urinary disorders such as urinary difficulty, excessive urination or incontinence
* Known overt bacterial infections in the skin;
* Known pregnancy;
* Known severe medical conditions, such as cardiovascular, liver or renal dysfunction or Diabetes Mellitus;
* Having used oral corticosteroids, oral antibiotics, other immunosuppressive or any preparation of oral herbal medicines for the treatment of AD in the past month;
* Having been diagnosed with scabies, allergic contact dermatitis, seborrheic dermatitis or psoriasis;
* Has taken anti-coagulant or anti-platelet drugs in the past month;
* Has taken any probiotics, prebiotics in the last month; and
* Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
EASI score | 12 weeks
  The change of EASI score for atopic dermatitis at week 12 Min value: 0, max value: 72, higher scores mean worse outcome. To assess the severity of atopic dermatitis.

SECONDARY OUTCOMES:
EASI score | 6 weeks
  The change of EASI score for atopic dermatitis at week 6 Min value: 0, max value: 72, higher scores mean worse outcome. To assess the severity of atopic dermatitis
EASI score | 16 weeks
  The change of EASI score for atopic dermatitis at week16 Min value: 0, max value: 72, higher scores mean worse outcome. To assess the severity of atopic dermatitis
CDLQI score | 12 weeks
  The change of CDLQI score at week 12 Min value: 0, max value: 30, higher scores mean worse outcome. To assess the quality of life of subjects.
CDLQI score | 16 weeks
  The change of CDLQI score at week 16 Min value: 0, max value: 30, higher scores mean worse outcome. To assess the quality of life of subjects.
POEM score | 12 weeks
  The change of POEM score at week 12 Min value: 0, max value: 28, higher scores mean worse outcome. To assess the subjective symptoms of subjects.
POEM score | 16 weeks
  The change of POEM score at week 16 Min value: 0, max value: 28, higher scores mean worse outcome. To assess the subjective symptoms of subjects.
Microbiome | 12 weeks
  The change of microbiome at week 12. The oral and gut microbiota are the collection of microbial agents such as bacteria, viruses and fungi that inhabit in the mouth cavity and gut. Bacterial microbiome sequencing is performed using 16S ribosomal RNA pyrosequencing.
Time of flare | 16 weeks
  The time to reach flare (defined as major exacerbation disease increase > 50% of baseline EASI)
The number of subjects reaches flare | 16 weeks
  The number of subjects reaches flare (defined as major exacerbation disease increase > 50% of baseline EASI)
Trans-epidermal water loss (TEWL) | 6 weeks
  Trans-epidermal water loss (TEWL) at week 6 The Trans-epidermal water loss (TWEL) is measured in g/m2h, which range from 0 to 300. An increasing TEWL value indicates greater skin dryness.
Trans-epidermal water loss (TEWL) | 12 weeks
  Trans-epidermal water loss (TEWL) at week 12 The Trans-epidermal water loss (TWEL) is measured in g/m2h, which range from 0 to 300. An increasing TEWL value indicates greater skin dryness.
Trans-epidermal water loss (TEWL) | 16 weeks
  The change of trans-epidermal water loss (TEWL) at week 16 The TWEL is measured in g/m2h, which range from 0 to 300. An increasing TEWL value indicates greater skin dryness.
Skin hydration (SH) | 6 weeks
  The change of skin hydration (SH) at week 6 The SH is measured in arbitrary units (a.u.), which range from 0 to 300 a.u.
Skin hydration (SH) | 12 weeks
  The change of skin hydration (SH) at week 12 The SH is measured in arbitrary units (a.u.), which range from 0 to 300 a.u.
Skin hydration (SH) | 16 weeks
  The change of skin hydration (SH) at week 16 Skin hydration will be measured topically using the measuring device at a standard site below the antecubital fossa of each patient's right arm. The SH is measured in arbitrary units (a.u.), which range from 0 to 300 a.u.
Adverse event | 16 weeks
  Adverse event will be assessed in the study period

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Principal Investigator — Integrative Medical Centre
Locations (1):
- School of Chinese Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No